CLINICAL TRIAL: NCT07270172
Title: Multifactorial Intervention to Reduce Cardiac and Renal Oxygen Need in Type 1 Diabetes (the MICRON Study) - A Steno 1 Substudy
Brief Title: The MICRON Study - A Steno 1 Substudy
Acronym: MICRON
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: MICRON
Record Dates: First submitted 2025-11-14; First posted 2025-12-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetic Kidney Disease; Diabetes-Related Complications; Renal oxygenation; Cardiac oxygenation; Renal inflammation; Renal fibrosis; Cardiovascular disease
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Nephropathies; Diabetes Complications; Nephritis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (whole blood and plasma) Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group in the Steno 1 study: Receiving the intensive treatment therapy in the Steno 1 Study. This consists of more ambitious blood pressure and lipid targets as well as individualised pharmacological intervention with GLP1 receptor agonist (semglutide), dual SGLT-1/2 inhibitor (sotagliflozin), and/or nonsteroidal mineralocorticoid receptor antagonist (finerenone).
- Control group in the Steno 1 study.: Receiving standart care in the Steno 1 Study.

SUMMARY:
The goal of this observational study is to compare cardiac and renal oxygen consumption among subjects with type 1 diabetes treated with either multifactorial intervention or according to the current standard care. Participants are recruited from a main study /the Steno1 study) responsible for the intervention.

The main questions it aims to answer are if a multifactorial intervention in subjects with type 1 diabetes targeting cardiovascular and renal risk factors, will reduce cardiac and renal oxygen demand.

Participants will undergo the following examinations at 0-month, 6-month, and 24-month after enrolling in the main study:

* Measurement of cardiac and real oxygen consumption ([11C]acetate PET/CT-scan)
* Measurement of kidney function ([99mTc]DTPA GFR measurement)
* Measurement of markers of heart and kidney disease in blood and urine samples.

DETAILED DESCRIPTION:
In the MICRON study we will recruit participants from the ongoing CTIS approved Steno 1 study which is a prospective, cluster-randomized multicentre trial of 2000 persons with T1D. The Steno 1 study evaluates cardiovascular and renal effects of a multifactorial intervention vs. standard clinical care in subjects with type 1 diabetes (T1D) and established diabetic kidney disease (DKD), cardiovascular disease (CVD), heart failure, obesity or a >10% 5-year CVD risk using the Steno Risk Engine. The multifactorial intervention includes ambitious blood pressure and lipid targets as well as individualised pharmacological intervention with semglutide, sotagliflozin, and/or finerenone.

For the MICRON study we will recruit 20 persons from the ongoing Steno 1 study receiving multifactorial intervention as well as 20 persons from the Steno 1 study receiving standard care. No additional intervention is used for the MICRON study.

In the MICRON study each participant will undergo both [¹¹C]acetate PET/CT and [⁹⁹mTc]DTPAGFR measurements at baseline (inclusion) and again after 6 and 24 months of treatment (multifactorial intervention vs. standard care). At each of the three visits, blood and urine samples will be collected, along with anthropometric measurements.

The primary outcome variables, myocardial and renal oxygen consumption, will be assessed using [¹¹C]acetate PET/CT using a long axial field-of-view (LAFOV) PET scanner. Given that renal oxygen consumption is influenced by glomerular filtration rate (GFR), we will use [⁹⁹mTc]DTPA to accurately measure and account for variations in GFR when assessing renal oxygen consumption.

Three additional work packages WP2, WP3 and WP4 are to be conducted in collaboration with Steno Diabetes Centre Copenhagen, Monash University, Melbourne, Australia and the Department of Biomedicine, Aarhus University, Aarhus, Denmark investigating: WP2 Fibrosis, WP3 Oxidative stress and inflammation and WP4 Urinary extracellular vesicle proteomics.

ELIGIBILITY:
Steno 1 inclusion criteria:

* Male or female persons ≥40 years old with T1D (diagnosis before age 30 with insulin from onset or if diagnosis after 30 years of age insulin from onset and DKA or positive autoantibodies (in accordance with local guidelines), or confirmed, at the investigator's discretion by the available medical records) during >10 years.
* Presence of chronic kidney disease (UACR >30 mg/g or eGFR < 60 ml/min/1.73 m2) OR history of ischemic heart disease (previous myocardial infarction, stroke or angina) OR history of heart failure OR obesity grade 2 and 3 (BMI>35 kg/m2) OR 5-year CVD risk >10% according to Steno Type 1 Risk Engine.
* Fertile females must use highly efficient chemical, hormonal and mechanical contraceptives during the whole study and at least 2 months after cessation of study drug. The following contraceptive methods are approved: IUD or hormonal contraception that inhibits ovulation, i.e. pills, implantations, transdermal patches, vaginal ring or depot injection. Alternatively, be in menopause (i.e. must not have had regular menstrual bleeding for at least one year), have undergone bilateral oophorectomy or have been surgically sterilized or hysterectomised at least 12 months prior to screening.
* Ability to communicate with the investigator and understand informed consent.
* Given written informed consent.

Steno 1 exclusion criteria:

* Type 2 Diabetes, Maturity-onset diabetes of the young (MODY), secondary diabetes.
* History of pancreatitis.
* Body mass index < 18.5 kg/m2
* Females of childbearing potential who are pregnant, breast-feeding, intend to become pregnant or are not using adequate contraceptive methods.
* Known or suspected abuse of alcohol or recreational drugs.
* Participant in another drug-intervention study.
* Chronic Kidney Disease stage 5.

Additional exclusion criteria in the MICRON study:

* Active malignant disease
* Use of study drugs (SGLT inhibitors, GLP-1 RA, or finererone) at inclusion.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for the Steno1 Study is persons with Type 1 Diabetes at the Steno Diabetes Centre and at partner clinics in Region Midt, Denmark. The MICRON study will recruit from these participants.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Myocardial oxygen consumption | At baseline (0 month), at 6 months and 24 months.
  Measured by [11C]acetate PET/CT Unit: volumen pr mass pr time
Renal oxygen consumption | At baseline (0 month), at 6 months and 24 months.
  Measured by [11C]acetate PET/CT Unit: volumen pr mass pr time

SECONDARY OUTCOMES:
Myocardial external efficiency | At baseline (0 month), at 6 months and 24 months.
  Measured by [11C]acetate PET/CT Unit: %
Myocardial perfusion | At baseline (0 month), at 6 months and 24 month.
  Measured by [11C]acetate PET/CT Unit: volumen pr mass pr time
Renal perfusion | At baseline (0 month), at 6 months and 24 months.
  Measured by [11C]acetate PET/CT Unit: volumen pr mass pr time
Amount of markers for oxidative stress and inflammation | Samples collected at baseline (0 month), at 6 months and 24 months.
  Exploratory analysis on pathways of oxidative stress and inflammation known to be involved in diabetic cardiorenal damage. Analysis on blood and urine samples.
Amount of markers for renal fibrosis | Samples collected at baseline (0 month), at 6 months and 24 months.
  Exploratory measurements of renal extracellular matrix metabolism. Measurement of formation of collagen type III and VI (PRO-C3 and PRO-C6), endotrophin, and the collagen III degradation product C3M in blood and urine.
Urinary extracellular vesicle | On urine samples collected at baseline (0 month), at 6 months and 24 months. Differential protein abundance is assessed longitudinally (baseline vs 6 and 24 months) and cross-sectionally between treatments at matched time points.
  Unbiased, large-scale quantitative proteomic profiling of urinary extracellular vesicles (uEVs). Functional interpretation uses Gene Ontology and pathway enrichment analyses, with emphasis on inflammation, mitochondrial oxygen consumption, and oxidative-stress-related pathways.
Glomerular filtration rate | At baseline (0 month), at 6 months and 24 months.
  Measured by [99mTc]DTPA Unit: ml/(min*1,73 m^2)
Urine albumin-creatinine ratio | At baseline (0 month), at 6 months and 24 months. Moreover, results from in-clinic laboratory assessments will be collected during the study period if available.
  Measured by urine spots Unit: None

OTHER OUTCOMES:
Blood pressure | At baseline (0 month), at 6 months and 24 months.
  Unit: mmHg
Plasma glucose | Will be measured regularly (at least hourly) at the three study visits (baseline, 6 months, and 24 months) to monitor levels during fasting.
  Measured by POCT (Point-of-Care Testing)
Pro-brain natriuretic peptide | At baseline (0 month), at 6 months and 24 months.
  Unit: Mass pr volumen
Troponin I | At baseline (0 month), at 6 months and 24 months.
  Unit: Mass pr volumen
Blood lipids | At baseline (0 month), at 6 months and 24 months.
  Total cholesterol, LDL, HDL and triglycerides. Unit: Mass pr volumen
Liver enzymes | At baseline (0 month), at 6 months and 24 months.
  Alanine transaminase (ALAT) and aspartate transaminase (ASAT). Unit: Mass pr volumen.
Hemoglobin A1c | At baseline (0 month), at 6 months and 24 months.
  Unit: mmol/mol
Thyroid-stimulating hormone (TSH) | At baseline (0 month), at 6 months and 24 months.
  Unit: amount pr volumen.
Blood ketones | At baseline (0 month), at 6 months and 24 months.
  Unit: amount per volumen
eGFR | At baseline (0 month), at 6 months and 24 months.
  Unit: mL/min/1,73 m2
Electrolytes | At baseline (0 month), at 6 months and 24 months.
  Sodium + Potassium Unit: mass pr
Trombocytes | At baseline (0 month), at 6 months and 24 months.
  Unit: amount pr volumen.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob A Østergaard, MD, PhD, Principal Investigator — Steno Diabetes Centre Aarhus
Locations (5):
- Denmark (5):
  - Aarhus University Hospital, Aarhus N
  - Regionshospitalet Gødstrup, Gødstrup
  - Regionshospitalet Horsens, Horsens
  - Regionshospitalet Silkeborg, Silkeborg
  - Regionshospitalet Vibrg, Viborg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Stougaard EB, Andersen MR, Bagger JI, Sondergaard E, Ostergaard JA, Curovic VR, Persson F, Almdal T, Mathiesen AS, Andries A, Bohl M, Norgaard LJ, Dejgaard TF, Dorfinger GH, Gustenhoff P, Gaede PH, Hamid YH, Johannesen HL, Juhl CB, Jorgensen ME, Kielgast U, Kofoed-Enevoldsen A, Lindhardt M, Mortensen LS, Thomsen HH, Stidsen J, Sorensen LP, Urhammer S, Rossing P; Steno 1 Study Group. The Steno 1 study: Multifactorial intervention to reduce cardiovascular disease in type 1 diabetes-rationale and protocol of the prospective, randomized, open-labelled multicentre study. Diabetes Obes Metab. 2025 Oct;27(10):5432-5443. doi: 10.1111/dom.16606. Epub 2025 Jul 29. PMID 40726451